CLINICAL TRIAL: NCT06989554
Title: Efficacy of a Low-Cost Tactile Incentiviser for Improving Partial Weight-Bearing Accuracy During Early Inpatient Rehabilitation After Lower-Limb Surgery: A Single-Centre Pilot Randomised Controlled Trial
Brief Title: Tactile Incentiviser Improves Partial Weight Bearing After Lower-Limb Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi dell'Insubria (Other)
Responsible Party: Principal Investigator, Piero Antonio Zecca, Researcher, Università degli Studi dell'Insubria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 026262
Record Dates: First submitted 2025-05-07; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Femoral Fractures; Pelvic Fractures; Hip Fractures (ICD-10 72.01-72.2); Hip Arthroplasty; Knee Arthroplasty; Ankle Fractures
Keywords: partial weight bearing; tactile biofeedback insole; load-monitoring device; postoperative gait training; orthopaedic rehabilitation; lower-limb surgery; hip replacement rehab; femoral shaft fixation; pressure sensor calibration; System Usability Scale (SUS)
MeSH Terms: conditions — Femoral Fractures; Hip Fractures; Ankle Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentivator (Experimental): Participants received a calibrated rubber insole containing four spring-loaded snap buttons that collapse and provide an immediate plantar tactile cue whenever the load on the operated limb exceeds 20 % ± 1 % of body weight. The insole was fitted on postoperative day 1 and worn inside the surgical-side shoe during every supervised ambulation session (walker or crutches) until hospital discharge (≈ 14 days, median 6 sessions per day). Patients were instructed to unload the limb instantly whenever the tactile "click" was felt. No batteries, electronics or external displays were used; calibration was performed once on a hydraulic press before first use.
  Interventions: Device: mechanical feedback insole
- Standard Physiotherapy (Active Comparator): Participants received routine ward physiotherapy only. Verbal instructions and a single bathroom-scale drill were used to teach 20 % body-weight partial loading, but no insole, sensor or tactile feedback device was provided thereafter. Treatment frequency, walking aids, pain management and discharge criteria were identical to the intervention arm.
  Interventions: Procedure: Standard physiotherapy without feedback device

INTERVENTIONS:
Device: mechanical feedback insole — A 3-mm rubber insole containing four 15-mm spring-steel snap buttons aligned along the heel-mid-foot axis. Each insole is statically calibrated on a hydraulic press so that the buttons collapse at 20 % ± 1 % of the individual's body weight, producing an unmistakable plantar cue when the load limit is exceeded. The device is purely mechanical, requires no batteries, and is fitted on postoperative day 1. Participants wear the insole during every supervised walking session until discharge (≈ 14 days).
  Arms: Incentivator
Procedure: Standard physiotherapy without feedback device — Routine inpatient physiotherapy consisting of verbal instruction to limit loading to 20 % body weight, initial bathroom-scale training, and assisted ambulation with walker or crutches. No tactile, visual, or electronic feedback device is provided. Session frequency, walking aids, analgesia, and discharge criteria are identical to the intervention arm; duration ≈ 14 days.
  Arms: Standard Physiotherapy

SUMMARY:
Background: After lower-limb surgery, many patients are instructed to walk with only a fraction of their body weight on the operated leg (partial weight bearing). Traditional teaching methods-verbal instructions or brief practice with a bathroom scale-often fail to maintain the load within a safe range, potentially increasing the risk of delayed bone healing or implant failure.

Purpose: This pilot study investigates whether a very low-cost, purely mechanical "tactile incentiviser" placed inside the shoe can assist participants in adhering to a 20% body-weight limit during the first two weeks of inpatient rehabilitation.

Design: Single-centre, parallel-group, randomised controlled trial. Thirty-four adults undergoing hip or knee arthroplasty, or surgery for femoral-shaft or pelvic fracture, were enrolled. Randomisation was performed using a computer-generated list in sealed envelopes. Outcome assessors were blinded.

Intervention: The device consists of four spring buttons embedded in a rubber insole that collapse and deliver a tactile cue when the 20% ± 1% load threshold is exceeded. Participants in the intervention group wore the insole during supervised walking sessions. Control participants received standard physiotherapy without feedback devices.

Primary Outcome: Absolute deviation (kg) between prescribed and actual load, assessed with a pressure sensor at baseline and discharge.

Secondary Outcomes: Pain intensity (NRS), Six-Minute Walk Test (6MWT) distance, and usability (System Usability Scale, SUS).

Note: No results or conclusions are included here. Results will be reported in the appropriate Results Section after the study is completed.

DETAILED DESCRIPTION:
Background and Rationale Partial weight-bearing (PWB) restrictions (10-30% of body weight) are routinely prescribed for 2-6 weeks following hip or knee arthroplasty, fracture fixation, and pelvic or ankle reconstruction. Failure to adhere to these limits may overload internal fixation devices, delay bone healing, or impair implant osseointegration. While electronic smart-insole systems can enhance load accuracy, they often cost over €600, require batteries and smartphone connectivity, and are not readily available in low-resource settings. Therefore, a purely mechanical "tactile incentiviser" was developed to provide an immediate plantar cue when the load threshold is exceeded, aiming to offer a low-cost alternative.

Device Design and Calibration The incentiviser has a 3-mm rubber insole incorporating four spring-steel snap-buttons (15 mm diameter, 4 mm height) aligned along the heel-midfoot axis. Three interchangeable polyurethane-foam pads (35 / 45 / 60 Shore A, 6 mm thickness) allow adjustment according to participant body mass. Each insole is statically calibrated using a custom hydraulic press with a 0-500 N load cell (accuracy ± 0.5 N), increasing in 10 N increments until the buttons collapse at a target of 20% ± 1% of body weight. Calibration is performed in triplicate to ensure repeatability.

Study Design This is a single-centre, assessor-blinded, parallel-group pilot randomised controlled trial. Ethical approval was granted by the Institutional Review Board of the University of Insubria (protocol number 0026262).

Participants Eligible participants are adults aged 18-85 years undergoing hip or knee arthroplasty, femoral-shaft fracture intramedullary nailing, or pelvic fracture fixation who can ambulate ≥ 5 meters with assistive devices. Exclusion criteria include neurological gait disorders, pre-existing non-weight-bearing status, and foot sizes outside the 35-47 EU range.

Randomisation and Allocation Concealment All eligible admissions are listed chronologically each calendar week and assigned an incremental study ID. An independent researcher uses Random.org to randomly allocate three participants to the intervention arm and three to the control arm via simple random sampling without replacement. The allocation list is disclosed to ward staff only after baseline assessment to maintain allocation concealment. Outcome assessors and data analysts are blinded to group assignment. Due to the nature of the intervention, participants and therapists are not blinded.

Interventions Intervention Arm: Participants wear the calibrated incentiviser in the surgical-side shoe during every supervised walk starting from post-operative day 1 until discharge (approximately 14 days). Instructions are provided to encourage load reduction in response to the tactile cue.

Control Arm: Participants receive standard physiotherapy, including verbal instruction to limit loading to 20% of body weight and assisted practice using a walker or crutches, without any feedback device.

Outcome Measures Primary Outcome: Absolute deviation in kilograms from the prescribed 20% body weight load, measured using a validated wireless in-shoe pressure-sensor system (GeBioM-MobilData) during a 10-meter walk at baseline (T0) and at discharge (T1).

Secondary Outcomes: (i) Pain intensity using a 0-10 Numerical Rating Scale (NRS); (ii) Walking distance during the Six-Minute Walk Test (6MWT); (iii) Usability of the device assessed using the System Usability Scale (SUS) at T1.

Sample Size Justification A priori sample size calculation was based on an expected mean difference of 3 kg with a standard deviation of 5 kg, alpha = 0.05, and 80% power, yielding a required sample of 26 participants. The total sample was increased to 34 participants (17 per arm) to accommodate potential attrition.

Statistical Analysis Plan Between-group comparisons are planned using independent-samples t-tests (two-tailed, α = 0.05). Effect sizes will be reported using Cohen's d and corresponding 95% confidence intervals. Additional exploratory analyses will be conducted using two-way ANOVA, including diagnosis-stratified comparisons and interaction effects. All analyses will be performed using SPSS v19 and R v4.3.

Safety Monitoring The device is expected to be well tolerated, with no anticipated adverse effects. Skin condition will be monitored daily. Any adverse events will be recorded and reported to the IRB according to institutional guidelines.

ELIGIBILITY:
Inclusion Criteria:

Recent lower-limb orthopaedic surgery with a prescription of 20 % body-weight partial weight bearing: femoral-shaft fracture fixation, pelvic fracture fixation, total hip arthroplasty, hip hemi-arthroplasty, total knee arthroplasty, or trimalleolar ankle fracture fixation.

Able to stand and walk ≥ 5 m with a walking aid on postoperative day 1.

Sufficient cognitive capacity and language skills to follow instructions and provide written informed consent.

Exclusion Criteria:

Pre-existing gait disorder or neurological condition affecting load perception (e.g., stroke, Parkinson's disease, peripheral neuropathy, spinal cord injury).

Surgeon-ordered non-weight-bearing restriction.

Foot size < EU 35 or > EU 47, which cannot be accommodated by the insole.

Active foot ulcer, severe peripheral vascular disease, or local infection on the operated limb.

Clinically significant cognitive impairment (MMSE < 24) or language barrier precluding comprehension of study procedures.

Participation in another interventional study that could influence gait within the past 30 days.

Any medical condition that, in the investigator's judgement, contraindicates participation (e.g., unstable cardiopulmonary status, uncontrolled pain ≥ 7/10 NRS).

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Absolute deviation (kg) between prescribed 20 % body-weight load and actual load during gait | Post-operative day 1 (baseline) and hospital discharge (~14 days post-op)
  The in-shoe pressure-sensor system (GeBioM MobilData) records vertical ground-reaction force for each step over a 10-m walkway. Load on the operated limb is averaged across 20 consecutive steps. Deviation is calculated as the absolute difference (kg) between this value and the target 20 % of the patient's body weight. Lower scores indicate better adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Insubria, Varese, Varese, Italy

IPD SHARING:
Plan to Share IPD: No
ndividual-participant datasets will not be shared because the study is a single-centre pilot with a small sample size (n = 34) and contains potentially identifying gait-pressure traces. Only aggregate, de-identified results will be available in the published manuscript and ClinicalTrials.gov results section.

REFERENCES:
- [Background] Amoruso E, Dowdall L, Kollamkulam MT, Ukaegbu O, Kieliba P, Ng T, Dempsey-Jones H, Clode D, Makin TR. Intrinsic somatosensory feedback supports motor control and learning to operate artificial body parts. J Neural Eng. 2022 Jan 24;19(1):016006. doi: 10.1088/1741-2552/ac47d9. PMID 34983040
- [Background] Tamburella F, Lorusso M, Tagliamonte NL, Bentivoglio F, Bigioni A, Pisotta I, Lancini M, Pasinetti S, Ghidelli M, Masciullo M, Saraceni VM, Molinari M. Load Auditory Feedback Boosts Crutch Usage in Subjects With Central Nervous System Lesions: A Pilot Study. Front Neurol. 2021 Jul 6;12:700472. doi: 10.3389/fneur.2021.700472. eCollection 2021. PMID 34295303
- [Background] van Lieshout R, Pisters MF, Vanwanseele B, de Bie RA, Wouters EJ, Stukstette MJ. Biofeedback in Partial Weight Bearing: Usability of Two Different Devices from a Patient's and Physical Therapist's Perspective. PLoS One. 2016 Oct 31;11(10):e0165199. doi: 10.1371/journal.pone.0165199. eCollection 2016. PMID 27798674
- [Background] Hustedt JW, Blizzard DJ, Baumgaertner MR, Leslie MP, Grauer JN. Current advances in training orthopaedic patients to comply with partial weight-bearing instructions. Yale J Biol Med. 2012 Mar;85(1):119-25. Epub 2012 Mar 29. PMID 22461750